CLINICAL TRIAL: NCT04968431
Title: Three Dimensional Versus Two Dimensional Echocardiography in Assessment of Severity and Scoring of Rheumatic Mitral Stenosis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ibrahim Sayed, resident doctor, Assiut University
Other Study IDs: rheumatic mitral stenosis
Record Dates: First submitted 2021-06-16; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Mitral Valve Stenosis
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mitral Stenosis patient
  Interventions: Other: 2D Echocardiography; Other: 3D Echocardiography

INTERVENTIONS:
Other: 2D Echocardiography — Mitral valve area will be determined by 2 D echo-Doppler methods
Other: 3D Echocardiography — Patients included in the study will undergo 3D Echo after being evaluated with 2D Echo. Mitral valve area will be determined by real time 3D.

SUMMARY:
Although the prevalence of rheumatic fever is decreasing in developed countries, it still affects numerous areas in the non- industrialized world. Untreated mitral stenosis (MS) contributes significantly to global morbidity and mortality. Echocardiography is the main diagnostic imaging modality for evaluation of mitral valve (MV) obstruction and assessment of severity and hemodynamic consequences of MS as well as valve morphology. According to current guidelines and recommendations for clinical practice, the severity of MS should not be defined by a single value but assessed by valve areas, mean Doppler gradients, and pulmonary pressures. Transthoracic echocardiography is usually sufficient to grade MS severity and to define the morphology of the valve. Transesophageal echocardiography is used when the valve cannot be adequately assessed with transthoracic echocardiography and to exclude intracardiac thrombi before a percutaneous or surgical intervention. Three-dimensional transthoracic and transesophageal echocardiographic assessment provide more detailed physiological and morphological information. Current definitive treatment for severe MS involves percutaneous balloon mitral valvuloplasty (PMBV) or surgery. The effectiveness of PMBV is related to the etiology of MS, and certain anatomic characteristics tend to predict a more successful outcome for PMBV, whereas other MV structural findings might suggest balloon valvuloplasty to be less likely successful or even contraindicated. Does 3D echo can add more useful information over 2 D echo that could change treatment decision?

ELIGIBILITY:
Inclusion Criteria:

1. Patient age range from 18 years to 60 years.
2. Patient with isolated mitral stenosis (except those with mild mitral regurgitation and are candidate for PTMC by 2D Echo evaluation).
3. Patient with normal left ventricular EF
4. patient both in sinus rhythm or atrial fibrillation

Exclusion Criteria:

1. Age below 18 years or above 60 years.
2. Patient with another valve lesion or more than mild mitral regurgitation.
3. Patient with impaired cardiac function.
4. Mitral stenosis of other etiology than rheumatic origin

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Gender Based: Yes
Study Population: will be taken as a total coverage over a period of 1 year from patients attending Assiut University Heart Hospital outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
benefit of 3D echocardiography in mitral stenosis severity | 1 year
  The added benefit of 3D echocardiography over 2D echo in evaluation of rheumatic mitral stenosis severity with pressure gradient
benefit of 3D echocardiography in mitral stenosis scoring | 1 year
  The added benefit of 3D echocardiography over 2D echo in evaluation of rheumatic mitral stenosis score

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carapetis JR, Steer AC, Mulholland EK, Weber M. The global burden of group A streptococcal diseases. Lancet Infect Dis. 2005 Nov;5(11):685-94. doi: 10.1016/S1473-3099(05)70267-X. PMID 16253886
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Background] Lang RM, Badano LP, Tsang W, Adams DH, Agricola E, Buck T, Faletra FF, Franke A, Hung J, de Isla LP, Kamp O, Kasprzak JD, Lancellotti P, Marwick TH, McCulloch ML, Monaghan MJ, Nihoyannopoulos P, Pandian NG, Pellikka PA, Pepi M, Roberson DA, Shernan SK, Shirali GS, Sugeng L, Ten Cate FJ, Vannan MA, Zamorano JL, Zoghbi WA; American Society of Echocardiography; European Association of Echocardiography. EAE/ASE recommendations for image acquisition and display using three-dimensional echocardiography. Eur Heart J Cardiovasc Imaging. 2012 Jan;13(1):1-46. doi: 10.1093/ehjci/jer316. No abstract available. PMID 22275509
- [Background] Wunderlich NC, Beigel R, Siegel RJ. Management of mitral stenosis using 2D and 3D echo-Doppler imaging. JACC Cardiovasc Imaging. 2013 Nov;6(11):1191-205. doi: 10.1016/j.jcmg.2013.07.008. PMID 24229772